CLINICAL TRIAL: NCT05223049
Title: Evaluation of Neuropathic Pain in Patients With Psoriatic Arthritis
Brief Title: Neuropathic Pain in Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-06/95
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Psoriatic Arthritis
Keywords: Neuropathic Pain; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psoriatic Arthritis patients with neuropathic pain: Patients diagnosed with Psa according to The Classification Criteria for Psoriatic Arthritis (CASPAR) psoriatic arthritis criteria. Who has a DN4 score of ≥4 or PainDETECT score of ≥13.
  Interventions: Other: painDETECT questionnaire; Other: Douleur Neuropathique 4 questionnaire (DN4); Other: Short form-36; Other: Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC); Other: Numeric Rating Scale; Other: Disease activity in psoriatic arthritis (DAPSA)
- Psoriatic Arthritis patients with nonneuropathic pain: Patients diagnosed with Psa according to The Classification Criteria for Psoriatic Arthritis (CASPAR) psoriatic arthritis criteria. Who has a DN4 score of ≤4 or PainDETECT score of ≤13.
  Interventions: Other: painDETECT questionnaire; Other: Douleur Neuropathique 4 questionnaire (DN4); Other: Short form-36; Other: Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC); Other: Numeric Rating Scale; Other: Disease activity in psoriatic arthritis (DAPSA)

INTERVENTIONS:
Other: painDETECT questionnaire — The painDETECT questionnaire was specifically developed to detect neuropathic pain components in adult patients with low back pain. It is also used in detecting the neuropathic pain in rheumatic diseases. A score between ≤12 represents a nonneuropathic pain, ≥13 and ≤18 represents a possible neuropathic pain, while a score of ≥19 represents a neuropathic pain.
Other: Douleur Neuropathique 4 questionnaire (DN4) — DN4 is a clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient and 3 items based on the clinical examination. A score of ≥4 represents a neuropathic pain.
Other: Short form-36 — The 36-Item Short Form Survey (SF-36) is a self-reported measure of health. It comprises 36 questions which cover eight domains of health. 1) Limitations in physical activities because of health problems. 2) Limitations in social activities because of physical or emotional problems 3) Limitations in usual role activities because of physical health problems 4) Bodily pain 5) General mental health (psychological distress and well-being) 6) Limitations in usual role activities because of emotional problems 7) Vitality (energy and fatigue) 8) General health perceptions. Each domain is scored between 0 and 100 and a higher score represents a better outcome.
Other: Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC) — SPARCC was created as a measure for enthesitis in spondyloarthritis in general. It assesses 16 enthesial sites. Total number of the enthesitis is the total score of the evaluation. Total score is between 0 and 16, and higher scores represent a worse outcome.
Other: Numeric Rating Scale — Self reported pain scored between 0 (minimum)-10 (maximum). Higher scores represent a worse outcome.
Other: Disease activity in psoriatic arthritis (DAPSA) — DAPSA includes a 68/66 joint count summed with a patient global, patient pain score, and C- reactive protein level. The DAPSA provides a continuous score of arthritis activity and has validated cut points for remission (< 4) and low disease activity (< 14).

SUMMARY:
Pathogenesis of inflammatory diseases is suitable for eliciting neuropathic pain. The aim of this study is to evaluate the frequency of NP among PsA patients and relationship between disease activity, quality of life, functionality, and other numerous factors.

DETAILED DESCRIPTION:
Neuropathic pain (NP) is the pain arising from a primary lesion or a dysfunction of nervous system. NP can affect central or peripheral nervous system and can be caused by numerous factors such as inflammation or neuroplastic changes. Inflammation can sensitize nociceptors in sensory nerves by promoting prostaglandin E2 and I2 secretion thus, cause neuropathic pain. Besides, a mixed pain pattern with neuropathic components is thought to be developed in chronic pain conditions. In this point of view, pathogenesis of inflammatory diseases is suitable for eliciting NP. In arthritic joints, even non-arthritic tissues are affected by the disease and a condition called peripheral sensitization develops. Previous studies about NP and inflammatory diseases link have focused on rheumatoid arthritis and number of studies about NP and psoriatic arthritis (PsA) is limited. In this manner the aim of this study is to evaluate the frequency of NP among PsA patients and relationship between disease activity, quality of life, functionality, and other numerous factors.

ELIGIBILITY:
Inclusion Criteria:

* being aged≥18
* being diagnosed PSA according to CASPAR criteria

Exclusion Criteria:

* additional conditions that could cause neuropathic pain (e.g. radiculopathy, polyneuropathy, depression, fibromyalgia)
* history of fracture or surgery
* endocrinopathies that could cause neuropathic pain (e.g. DM)
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult psoriatic arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Frequency neuropathic pain in psoriatic arthritis patients | 1 day
  The frequency of neuropathic pain in the PSA patients included in the study according to painDETECT and DN4 scores.
Disease activity in Psoriatic arthritis (DAPSA) score in two groups | 1 day
  The statistical difference between two groups in terms of disease activity
Numeric Rating Scale (rest, movement) in two groups | 1 day
  The statistical difference between two groups in terms of disease activity
Short form-36 survey in two groups | 1 day
  The statistical difference between two groups in terms of SF-36 and subdomains
SPARCC enthesitis index in two groups | 1 day
  he statistical difference between two groups in terms of SPARCC

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] Ramjeeawon A, Choy E. Neuropathic-like pain in psoriatic arthritis: evidence of abnormal pain processing. Clin Rheumatol. 2019 Nov;38(11):3153-3159. doi: 10.1007/s10067-019-04656-5. Epub 2019 Jul 19. PMID 31325065